CLINICAL TRIAL: NCT00857831
Title: Vitamin D and Calcium Replacement/Supplementation in Subjects With Chronic Spinal Cord Injury
Brief Title: Vitamin D and Calcium Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B4162C-8
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; Vitamin D deficiency; Functional Electrical Stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Vitamin D Deficiency | interventions — Vitamin D; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Vitamin D & Calcium supplementation in FES
  Interventions: Dietary Supplement: Vitamin D and Calcium

INTERVENTIONS:
Dietary Supplement: Vitamin D and Calcium — 2000 IU/day Vitamin D3 (cholecalciferol) and 1.3 g/day calcium carbonate will be taken for 15-20 weeks.

SUMMARY:
Vitamin D aids in the body's ability to absorb calcium, it is a vital component in bone formation and break down. Reduced levels of vitamin D can indicate a vitamin deficiency and may depress serum calcium levels. The following is a list of common causes of vitamin D deficiency: lack of dairy products, alcohol usage, elderly, lack of exposure to sunlight, individuals with reduced mobility, GI malabsorption problems, dark complexion, severe liver damage, and renal failure. Many of these factors can be found in individuals with spinal cord injury. SCI results in disuse bone loss after acute injury, which continues with duration of injury. The goal of this study is to determine the effects of vitamin D and calcium supplements on calcium metabolism and vitamin D deficiency in individuals undergoing functional electrical stimulation (FES) stand retraining (SRT).

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury (paraplegia or quadriplegia)
* Vitamin D deficiency
* Absolute deficient Vitamin D [25(OH)D] < 16 ng/ml
* Relative deficient Vitamin D [25(OH)D] <30ng/ml - participation in the FES/SRT study at Kessler Institute for Rehabilitation

Exclusion Criteria:

* History of kidney stones
* History of bone disorders
* Currently pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Effects of Vitamin D and Calcium supplements on calcium metabolism and vitamin D deficiency | 15-20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Bauman, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States